CLINICAL TRIAL: NCT04363996
Title: Clinical Evaluation of New Bioactive Restorative Material Versus Resin Modified Glass Ionomer in Restoration of Cervical Lesions: Randomized Controlled Trial
Brief Title: Bioactive Restorative vs GIC Modified Glass Ionomer in Restoration of Cervical Lesions: Randomized Controlled Trial
Acronym: ActivaPresto
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amera Nabel, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1176
Record Dates: First submitted 2020-04-20; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Clinical Performance Using Modified USPHS Criteria

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- New Bioactive Restorative Material (Experimental): Activa Presto Bioactive restorative material
  Interventions: Other: New Bioactive Restorative Material
- Resin Modified Glass Ionomer (Active Comparator): Fuji II
  Interventions: Other: New Bioactive Restorative Material

INTERVENTIONS:
Other: New Bioactive Restorative Material — Filling material

SUMMARY:
Bioactive restorative materials are relatively new in dentistry. Activa BioACTIVE (Pulpdent Corporation, Watertown, MA) dual cured material is the first dental restoratives with a bioactive resin matrix, shock-absorbing resin component and reactive glass ionomer fillers designed to mimic the physical and chemical properties of natural teeth. It is a highly esthetic bioactive hydrophilic composite that bonds chemically to teeth, seals against 4 microleakage and releases more calcium, phosphate, and fluoride. It is delivered via a dualbarrel, automix syringe using a special dispensing gun. The company states that Activa is more bioactive than glass ionomers while more durable and fracture resistant than composites (ACTIVA BioACTIVE RESTORATIVE - Pulpdent).

DETAILED DESCRIPTION:
The resin composites used with bonding agents are popularly used for the restoration of cervical lesions. These materials exhibit high strength and physical properties as well as good esthetic property but they don't offer the chemical bonding and fluoride release potentials necessary for managing high caries risk patients (Khoroushi et al., 2012).

Fluorides containing restorative materials have been advocated as the material of choice for restoring cervical lesions in high caries risk patients since this kind of material offers chemical bonding, fluoride release, and caries inhibiting potentials. Conventional Glass Ionomer and Resin modified glass ionomer restorative materials have high fluoride release and could be specified clinically to repair cervical lesions in high caries risk patients. However, clinical acceptance of these materials has been limited because of their low tensile strength, brittleness, and low resistance to wear (Somani et al., 2016).

Bioactive restorative materials are relatively new in dentistry. Activa BioACTIVE (Pulpdent Corporation, Watertown, MA) dual cured material is the first dental restoratives with a bioactive resin matrix, shock-absorbing resin component and reactive glass ionomer fillers designed to mimic the physical and chemical properties of natural teeth. It is a highly esthetic bioactive hydrophilic composite that bonds chemically to teeth, seals against 4 microleakage and releases more calcium, phosphate, and fluoride. It is delivered via a dualbarrel, automix syringe using a special dispensing gun. The company states that Activa is more bioactive than glass ionomers while more durable and fracture resistant than composites (ACTIVA BioACTIVE RESTORATIVE - Pulpdent). Activa Presto light-cured material from Pulpdent is the company's newest product that features biomimicry as Activa Bioactive dual-cured material. It is available in a 1.2 mL syringe for easy application, and no longer need for a special dispensing gun to apply the material. Consequently, placement of the resin is precise and highly adaptive to the cavity margins. It is highly radiopaque (250%), so it can be easily followed on radiographs.

There are eight esthetic shades: A1, A2, A3, A3.5, B1, BW and two new darker cervical shades A4 and A6 which can be useful in geriatric patients. The material diffuses fluoride, calcium and phosphate ions that fortify the saliva and help replace essential minerals that are lost in the decay process. This highly esthetic light-cured resin contains these ions in a stackable resin matrix that holds its shape and does not slump. This durable product is resistant to fracturing and wear, especially so on the thin areas of enamel bevels, and is indicated for all restorative procedures replacing dentin and/or enamel, anterior or posterior (ACTIVA Presto - Pulpdent).

ELIGIBILITY:
Inclusion Criteria:

1. Cervical carious lesions anterior teeth and premolars.
2. Age 20-40 years.

Exclusion Criteria:

1. Rampant caries.
2. Pregnancy.
3. Disabilities.
4. Oral Dryness.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Surface texture | 6 months
  ordinal Criteria Scoring system (ordinal)
Surface texture | 1 year
  ordinal

SECONDARY OUTCOMES:
Marginal adaptation | 6 months
  ordinal
Marginal adaptation | 1 year
  ordinal

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No